CLINICAL TRIAL: NCT03145714
Title: To Study the Effect of Sevoflurane and Propofol Versus Sevoflurane and Dexmedetomidine on Postoperative Cognitive Dysfunction
Brief Title: To Study the Effect of Sevoflurane and Propofol V Sevoflurane and Dexmedetomidine on Postoperative Cognitive Dysfunction
Acronym: POCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr Anita Kulkarni, Principal Investigator, Rajiv Gandhi Cancer Institute & Research Center, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RGCI&RC
Record Dates: First submitted 2017-03-07; First posted 2017-05-09 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: POCD; Elderly
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol/Sevoflurane (Group P) (Experimental): Standard technique of induction of anaesthesia .
  Maintenance of anesthesia with intravenous (IV) Propofol Infusion at rate 100-150 mcg/kilogram/hour and Inhalational Anesthetic Sevoflurane during the surgery. Intervention is to titrate dosage of Propofol and Sevoflurane to maintain Bispectral Index between 40-60.
  Total dosage of IV Propofol and Sevoflurane uptake will be calculated at the end of surgery.
  Interventions: Drug: Maintainance of anesthesia with Intravenous Propofol infusion
- Dexmedetomidine/Sevoflurane (Group D) (Active Comparator): Standard technique of induction of anaesthesia .
  Maintenance of anesthesia with intravenous Dexmedetomidine Infusion at rate 1- 4 mcg/kilogram/hour and Inhalational Anesthetic Sevoflurane during the surgery.
  Intervention is to titrate dosage of Dexmedetomidine and Sevoflurane to maintain Bispectral Index between 40 - 60.
  Total dosage of IV Dexmedetomidine and Sevoflurane uptake will be calculated at the end of surgery.
  Interventions: Drug: Maintainance of anesthesia with Intravenous Dexmedetomidine

INTERVENTIONS:
Drug: Maintainance of anesthesia with Intravenous Propofol infusion — The dosage of Intravenous Propofol will be titrated to maintain BIS Values between 40 -60.
  Arms: Propofol/Sevoflurane (Group P)
Drug: Maintainance of anesthesia with Intravenous Dexmedetomidine — The dosage of Intravenous Dexmedetomidine will be titrated to maintain BIS Values between 40 -60.
  Arms: Dexmedetomidine/Sevoflurane (Group D)

SUMMARY:
Postoperative Cognitive Dysfunction (POCD), is a subtle decline in cognitive function characterized by impairment of memory and reduced ability to concentrate in elderly patients exposed to general anaesthesia. This prospective study aims to compare incidence and severity of POCD in two groups of patients. Group P receiving Intravenous Propofol and Inhalational anesthetic Sevoflurane. Group D receiving Intravenous Dexmedetomidine and Inhalational anesthetic Sevoflurane, Neuropsychological Test will be performed 24 hours before surgery and on postoperative day 3 and day 7.

DETAILED DESCRIPTION:
The adult patients posted for major surgery under general anesthesia will be included in the study, patients will be allotted randomly to either Group P (Propofol) or Group D (Dexmedetomidine). In the Operation Room (OR) monitoring Electrocardiography (ECG), Pulse Oximetry (SPO2), Noninvasive Blood Pressure (NIBP), End tidal Carbon di oxide (ETCO2) and Bispectral Index (BIS) Covidien, will be attached to all patients. In both groups Anesthesia will be induced with Fentanyl 1mcg /kg-1, Morphine 0.1mg/kg-1, Propofol 1-1.5mg /kg1- and neuromuscular blocking agent Atracurium 0.5 mg/kg-1. Oral Cuffed Endotracheal Tube (ETT) will be placed in the trachea. Anaesthesia will be maintained controlled ventilation , intermittent fentanyl boluses 20 mcg and in Group P with medicated Air/Oxygen (O2) with Fractional Inspired Oxygen (FiO2 50%), Sevoflurane and Propofol Infusion to maintain BIS between 40-60. In Group D anesthesia will be maintained with Medicated Air/Oxygen (FiO2 50%), Sevoflurane and Dexmedetomidine infusion to maintain BIS between 40-60. Intraoperatively monitoring of vitals, BIS numerical value, Minimum Alveolar Concentration (MAC) Value for Sevoflurane, Expired concentration of Sevoflurane and rate of infusion of Propofol/Dexmedetomidine will be noted every 30 minutes. Intraoperative decrease in Mean Arterial Pressure (MAP) < 60 mmHg, Heart rate (HR) < 50, SPO2 < 90 % will also be noted. At the end of surgery total dosage of Propofol/Dexmedetomidine and total amount of Sevoflurane consumed will be calculated. At the end of surgery neuromuscular blockade will be reversed. Total Duration of anesthesia will be noted. On emergence from anesthesia any episode of acute delirium will be recorded. Time from end of anesthesia to eye opening will be noted in both the groups. Neuropsychological Test consisting of Letter Digit Substitution Test, Trail Making Test Part A, Part B, Stroop Colour Word Test, Visual Verbal Learning Test will be performed 24 hours prior to surgery in the preanesthesia clinic and on postoperative day 3 and day 7.

ELIGIBILITY:
Inclusion Criteria:

* Patient subjected to general anaesthesia for elective noncardiac surgical procedure with duration above 2 hours and postoperative stay for 3 days. Patient should be available for follow up on 7 th postoperative day.

Exclusion Criteria:

* Patients having severe psychosis on antidepressant medications, cerebral disease, pre-existing cognitive dysfunction with Mini Mental State Examination (MMSE) Score less than 23, history of drug abuse, significant visual and hearing impairment ,language difficulties and illiteracy.

Ages: 58 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Postoperative Cognitive Dysfunction (POCD) after major noncardiac surgery under general anesthesia in Propofol and Dexmedetomidine Group | day 3 to day 7
  Postoperative Changes in Neuropsychological Tests Score compared with baseline preoperative Neuropsychological Test scores in both the groups.

SECONDARY OUTCOMES:
Recovery time from the stopping of anesthetics agents to eye opening in both Propofol and Dexmedetomidine Group | 30 seconds to 30 minutes.
  Time in seconds required for patients to respond to verbal commands on stopping the anesthetic agents in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kulkarni, M.D., Principal Investigator — Rajiv Gandhi Cancer Institue & Research Centre , Delhi, INDIA
Locations (2):
- India (2):
  - Dr Anita Kulkarni, Delhi
  - Rajiv Gandhi Cancer Institute and Research Centre, Delhi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deiner S, Silverstein JH. Postoperative delirium and cognitive dysfunction. Br J Anaesth. 2009 Dec;103 Suppl 1(Suppl 1):i41-46. doi: 10.1093/bja/aep291. PMID 20007989
- [Background] Akeju O, Pavone KJ, Westover MB, Vazquez R, Prerau MJ, Harrell PG, Hartnack KE, Rhee J, Sampson AL, Habeeb K, Gao L, Pierce ET, Walsh JL, Brown EN, Purdon PL. A comparison of propofol- and dexmedetomidine-induced electroencephalogram dynamics using spectral and coherence analysis. Anesthesiology. 2014 Nov;121(5):978-89. doi: 10.1097/ALN.0000000000000419. PMID 25187999
- [Background] Kotekar N, Kuruvilla CS, Murthy V. Post-operative cognitive dysfunction in the elderly: A prospective clinical study. Indian J Anaesth. 2014 May;58(3):263-8. doi: 10.4103/0019-5049.135034. PMID 25024467